CLINICAL TRIAL: NCT03285932
Title: Evaluation of Stereotactic Radiotherapy of the Resection Cavity After Surgery of Brain Metastases Compared to Post-operative Whole-brain Radiotherapy
Brief Title: Stereotactic Radiotherapy of the Resection Cavity of Brain Metastases vs. Post-operative Whole-brain Radiotherapy
Acronym: ESTRON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Juergen Debus (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Sponsor-Investigator, Juergen Debus, Prof. Dr. Dr. Jürgen Debus, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESTRON
Record Dates: First submitted 2017-09-13; First posted 2017-09-18 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Brain Metastases, Adult
Keywords: Brain Metastase; Radiation of resection cavity; WBRT (whole brain radiotherapy); SRS (stereotactic radiosurgery)
MeSH Terms: conditions — Brain Neoplasms; Snyder Robinson syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-operative SRS of resection cavity (Experimental): High-resolution contrast-enhanced post-operative MRI imaging in preparation for Cyberknife SRS. Cyberknife SRS of the resection cavity and all potential additional metastases diagnosed in the treatment planning MRI (up to 10 lesions)
  Resection cavity:
  7 x 5 Gy @ 95%-isodose
  Potential additional brain metastases:
  20 Gy @ 70%-isodose (lesions < 2 cm max. diameter) 18 Gy @ 70%-isodose (lesions 2 - 3 cm max. diameter) 6 x 5 Gy @ 70%-isodose (lesions > 3 cm max. diameter)
  Interventions: Radiation: post-operative stereotactic radiosurgery (SRS)
- Post-operative WBRT (Other): Post-operative WBRT will be performed according to the following dose regimen: 10 x 3 Gy
  Interventions: Radiation: Whole brain radiotherapy (WBRT)

INTERVENTIONS:
Radiation: post-operative stereotactic radiosurgery (SRS) — For radiosurgery, patients will be immobilized. Treatment planning including the MRI and planning CT should be performed 1 -2 weeks before SRT and treatment finished at latest 3-4 weeks after surgery. Planning should be as close to SRT as possible.
  Organs at risk such as the brain stem, optic nerves, chiasm and spinal cord will be contoured. The Clinical Target Volume 1 (CTV1) will be defined as the resection cavity based on MRI and CT including T1 contrast enhanced changes around the resection cavity. The Clinical Target Volume 2 (CTV2) will be defined as a 3mm margin added to CTV1 by isotropic expansion and slightly adjusted as deemed appropriated by the experienced contouring physician. The Planning Target Volume (PTV) will be an additional margin of 1mm added to CTV2 by isotropic expansion.
  Treatment planning will be performed using Accuray's Multiplan or subsequent approved treatment planning systems for Cyberknife.
  Arms: Post-operative SRS of resection cavity
Radiation: Whole brain radiotherapy (WBRT) — For WBRT, an individual head fixation mask is manufactured for each patient, and treatment planning is performed as virtual simulation or 3D-conformal RT planning based on CT-imaging. The portals include the whole brain with special focus as including the skull base areas and lamina cribrosa. For low infratentorial lesions, the treatment volume may include the whole brain down to the second cervical vertbra.
  RT will be applied with two portals (e.g. 87°and 273°) using a 6 MeV linear accelerator.
  For WBRT, a total dose of 30 Gy in 3 Gy fractions will be applied.
  Arms: Post-operative WBRT

SUMMARY:
In advanced cancer disease brain metastases are common, difficult to treat, and are associated with a poor prognosis. As new local and systemic therapies are eventually resulting in improved survival and quality of life for patients with brain metastases, negative neurocognitive effects of radiation therapy are becoming increasingly important as well as good loco-regional disease control of brain metastases.

Concerning treatment, brain metastases remain a major clinical problem and a multidisciplinary approach to management should be adopted. Neurosurgical resection with postoperative whole brain radiotherapy (WBRT) is one major treatment option in solitary or symptomatic brain metastases. Furthermore, WBRT is recommended for multiple brain metastases. For a limited number of brain metastases stereotactic radiosurgery (SRS) has been established as a highly effective treatment alternative.

Recently, a new treatment approach combing neurosurgery with postoperative stereotactic radiotherapy (SRT) of the resection cavity is emerging. Based on available evidence, postoperative SRT of the resection cavity improves local control following surgery, reduces the number of patients who require whole brain radiotherapy, and is well tolerated (1).

This protocol is aimed at primarily evaluating the safety and toxicity profile of SRT to the resection cavity following neurosurgical resection combined with SRT of potentially further unresected brain metastases, compared to postoperative whole-brain radiotherapy (WBRT). Secondary, the local effect of SRT in patients with brain metastases will be assessed by measuring time to local recurrence (LR), local and loco-regional progression-free survival (PFS).

Additional systemic treatment will be carried out according to the standards of the National Center for Tumor Therapy (NCT).

DETAILED DESCRIPTION:
Scientific Background: Brain metastases (BM) represent a significant healthcare problem. It is estimated that 20% to 40% of patients with cancer will develop metastatic cancer to the brain during the course of their illness 1. The most common primary sites are lung, melanoma, renal, breast and colorectal cancer 2. Options for patients with brain metastases had been limited to whole brain radiotherapy (WBRT) or supportive care alone, and systemic chemotherapy was often discontinued. Historically, the best possible supportive care or whole-brain radiotherapy (WBRT) were the standard of care 1 aiming at temporary symptom relief. For WBRT, efficacy in symptom relief but also in prolongation of the median survival time by 3-6 months is well documented. To date, microsurgical approaches and SRS, both proved to be safe and efficient, offer alternative treatment options that potentially meet these concerns 6,7. After proving its efficacy in achieving local tumor control in the treated volume, SRS was used as a stand-alone treatment option in patients with oligometastases (one to four metastases) in the brain. There is a rapidly expanding recent body of literature on outcomes of single-fraction SRS or hypofractionated SRS targeting the resection cavity after surgical resection of BM. Several retrospective series assessed the efficacy and safety of postoperative SRS to the resection cavity 9 aiming at an enhanced local tumor control but also at avoidance of the neurotoxic late effects of WBRT. WBRT followed by SRS of the tumor bed leads to 1-year local control rates of 70-93 %, which is comparable to results after surgery followed by WBRT. Median survival was 12-18 months with a 1-year incidence of new metastases in the brain of 45-60 %.

Trial Objectives: This protocol is primarily aimed at evaluating the safety and toxicity profile of SRS following neurosurgical resection and compares it to that of WBRT as the established standard of care. Secondary, the local effect of radiation therapy in patients with brain metastases will be assessed by measuring time to local and loco-regional recurrence, local and loco-regional PFS and overall survival at 12 months after treatment.

Patients´Selection: Patients with the diagnosis of brain metastases from solid tumors that have undergone neurosurgical resection of one brain metastasis will be evaluated and screened for the protocol. All patients fulfilling the inclusion and exclusion criteria will be informed about the study and included into the study if they declare informed consent. Registration for the study must be performed before the start of RT.

Trial Design: The trial will be performed as a single-center two-armed prospective randomized Phase II study. Patients will be randomized into an experimental arm and a control arm. All patients will receive post-operative contrast-enhanced cranial MRI imaging and imaging will be assessed by a radiologist. All available MRI sequences, including SPACE will be taken into consideration for the definition of treatment target lesions. Patients for whom the post-operative MRI reveals more than 10 suspect intracranial lesions (all sequences taken into account) will not be included in the trial.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed solid cancer
* MRI confirmed cerebral metastases
* Neurosurgical resection of one cerebral metastasis
* age ≥ 18 years of age
* Karnofsky Performance Score >60
* for women with childbearing potential, (and men) adequate contraception.
* ability to understand character and individual consequences of the clinical trial
* written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* refusal of the patients to take part in the study
* previous radiotherapy to the brain
* > 10 unresected brain metastases in postoperative MRI
* Patients who have not yet recovered from acute toxicities of prior therapies
* known carcinoma < 2 years ago (excluding carcinoma in situ of the cervix, basal cell carcinoma, squamous cell carcinoma of the skin) requiring immediate treatment interfering with study therapy
* pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
neurological progression-free survival (PFS) | 12 months PFS rate
  Neurologic progression-free survival in follow-up imaging is the primary endpoint of the study. The duration is defined as the time interval between the date start of RT and the date of local and loco-regional progression or death, or the date of leaving the study without local and loco-regional progression (e.g., lost to follow up non-local progression) whatever occurs first. Patients not reported local and loco-regional progressive or dead, or lost to follow-up or non-local progressive will be censored at the date of the last follow-up examination where no signs of local and loco-regional progression were observed.

SECONDARY OUTCOMES:
Overall survival (OS) | 12 months survival rate
  Time interval (days) between the date of RT begin and the date of death or date of leaving the study e.g., lost to follow up) whatever occurs first. Patients not reported dead or lost to follow-up will be censored at the date of the last follow-up or the time when last seen alive.
Local PFS | 12 months after treatment
  lenght of time (days) till local disease progression
Quality of life (QLQ-C30) | up to 12 months after treatment
  Units on a Scale
Loco-regional recurrence | up to 12 months after treatment
  Time to loco-regional recurrence
Quality of life (BN20) | up to 12 months after treatment
  Units on a Scale
Local recurrence | up to 12 months after treatment
  Time to local recurrence
Loco-regional PFS | 12 months after treatment
  lenght of time (days) till loco-regional disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Debus, Prof. Dr. Dr., Principal Investigator — Head of department Radiation Oncology
Locations (1):
- Department of Radiotherapy, University of Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsao MN, Lloyd N, Wong RK, Chow E, Rakovitch E, Laperriere N, Xu W, Sahgal A. Whole brain radiotherapy for the treatment of newly diagnosed multiple brain metastases. Cochrane Database Syst Rev. 2012 Apr 18;2012(4):CD003869. doi: 10.1002/14651858.CD003869.pub3. PMID 22513917
- [Background] Barnholtz-Sloan JS, Sloan AE, Davis FG, Vigneau FD, Lai P, Sawaya RE. Incidence proportions of brain metastases in patients diagnosed (1973 to 2001) in the Metropolitan Detroit Cancer Surveillance System. J Clin Oncol. 2004 Jul 15;22(14):2865-72. doi: 10.1200/JCO.2004.12.149. PMID 15254054
- [Background] Linskey ME, Andrews DW, Asher AL, Burri SH, Kondziolka D, Robinson PD, Ammirati M, Cobbs CS, Gaspar LE, Loeffler JS, McDermott M, Mehta MP, Mikkelsen T, Olson JJ, Paleologos NA, Patchell RA, Ryken TC, Kalkanis SN. The role of stereotactic radiosurgery in the management of patients with newly diagnosed brain metastases: a systematic review and evidence-based clinical practice guideline. J Neurooncol. 2010 Jan;96(1):45-68. doi: 10.1007/s11060-009-0073-4. Epub 2009 Dec 4. PMID 19960227
- [Background] Soliman H, Das S, Larson DA, Sahgal A. Stereotactic radiosurgery (SRS) in the modern management of patients with brain metastases. Oncotarget. 2016 Mar 15;7(11):12318-30. doi: 10.18632/oncotarget.7131. PMID 26848525
- [Background] Sperduto PW, Kased N, Roberge D, Xu Z, Shanley R, Luo X, Sneed PK, Chao ST, Weil RJ, Suh J, Bhatt A, Jensen AW, Brown PD, Shih HA, Kirkpatrick J, Gaspar LE, Fiveash JB, Chiang V, Knisely JP, Sperduto CM, Lin N, Mehta M. Summary report on the graded prognostic assessment: an accurate and facile diagnosis-specific tool to estimate survival for patients with brain metastases. J Clin Oncol. 2012 Feb 1;30(4):419-25. doi: 10.1200/JCO.2011.38.0527. Epub 2011 Dec 27. PMID 22203767
- [Background] Nieder C, Grosu AL, Gaspar LE. Stereotactic radiosurgery (SRS) for brain metastases: a systematic review. Radiat Oncol. 2014 Jul 12;9:155. doi: 10.1186/1748-717X-9-155. PMID 25016309
- [Background] Gans JH, Raper DM, Shah AH, Bregy A, Heros D, Lally BE, Morcos JJ, Heros RC, Komotar RJ. The role of radiosurgery to the tumor bed after resection of brain metastases. Neurosurgery. 2013 Mar;72(3):317-25; discussion 325-6. doi: 10.1227/NEU.0b013e31827fcd60. PMID 23208065
- [Background] Minniti G, Esposito V, Clarke E, Scaringi C, Lanzetta G, Salvati M, Raco A, Bozzao A, Maurizi Enrici R. Multidose stereotactic radiosurgery (9 Gy x 3) of the postoperative resection cavity for treatment of large brain metastases. Int J Radiat Oncol Biol Phys. 2013 Jul 15;86(4):623-9. doi: 10.1016/j.ijrobp.2013.03.037. Epub 2013 May 15. PMID 23683828
- [Background] Connolly EP, Mathew M, Tam M, King JV, Kunnakkat SD, Parker EC, Golfinos JG, Gruber ML, Narayana A. Involved field radiation therapy after surgical resection of solitary brain metastases--mature results. Neuro Oncol. 2013 May;15(5):589-94. doi: 10.1093/neuonc/nos328. Epub 2013 Mar 3. PMID 23460323
- [Background] Wang CC, Floyd SR, Chang CH, Warnke PC, Chio CC, Kasper EM, Mahadevan A, Wong ET, Chen CC. Cyberknife hypofractionated stereotactic radiosurgery (HSRS) of resection cavity after excision of large cerebral metastasis: efficacy and safety of an 800 cGy x 3 daily fractions regimen. J Neurooncol. 2012 Feb;106(3):601-10. doi: 10.1007/s11060-011-0697-z. Epub 2011 Aug 31. PMID 21879395
- [Background] Jensen CA, Chan MD, McCoy TP, Bourland JD, deGuzman AF, Ellis TL, Ekstrand KE, McMullen KP, Munley MT, Shaw EG, Urbanic JJ, Tatter SB. Cavity-directed radiosurgery as adjuvant therapy after resection of a brain metastasis. J Neurosurg. 2011 Jun;114(6):1585-91. doi: 10.3171/2010.11.JNS10939. Epub 2010 Dec 17. PMID 21166567
- [Background] Iorio-Morin C, Masson-Cote L, Ezahr Y, Blanchard J, Ebacher A, Mathieu D. Early Gamma Knife stereotactic radiosurgery to the tumor bed of resected brain metastasis for improved local control. J Neurosurg. 2014 Dec;121 Suppl:69-74. doi: 10.3171/2014.7.GKS141488. PMID 25434939
- [Background] Kelly PJ, Lin YB, Yu AY, Alexander BM, Hacker F, Marcus KJ, Weiss SE. Stereotactic irradiation of the postoperative resection cavity for brain metastasis: a frameless linear accelerator-based case series and review of the technique. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):95-101. doi: 10.1016/j.ijrobp.2010.10.043. Epub 2010 Dec 17. PMID 21168282
- [Background] Atalar B, Modlin LA, Choi CY, Adler JR, Gibbs IC, Chang SD, Harsh GR 4th, Li G, Nagpal S, Hanlon A, Soltys SG. Risk of leptomeningeal disease in patients treated with stereotactic radiosurgery targeting the postoperative resection cavity for brain metastases. Int J Radiat Oncol Biol Phys. 2013 Nov 15;87(4):713-8. doi: 10.1016/j.ijrobp.2013.07.034. Epub 2013 Sep 18. PMID 24054875
- [Background] Ojerholm E, Lee JY, Thawani JP, Miller D, O'Rourke DM, Dorsey JF, Geiger GA, Nagda S, Kolker JD, Lustig RA, Alonso-Basanta M. Stereotactic radiosurgery to the resection bed for intracranial metastases and risk of leptomeningeal carcinomatosis. J Neurosurg. 2014 Dec;121 Suppl:75-83. doi: 10.3171/2014.6.GKS14708. PMID 25434940
- [Background] Atalar B, Choi CY, Harsh GR 4th, Chang SD, Gibbs IC, Adler JR, Soltys SG. Cavity volume dynamics after resection of brain metastases and timing of postresection cavity stereotactic radiosurgery. Neurosurgery. 2013 Feb;72(2):180-5; discussion 185. doi: 10.1227/NEU.0b013e31827b99f3. PMID 23149969
- [Background] Jarvis LA, Simmons NE, Bellerive M, Erkmen K, Eskey CJ, Gladstone DJ, Hug EB, Roberts DW, Hartford AC. Tumor bed dynamics after surgical resection of brain metastases: implications for postoperative radiosurgery. Int J Radiat Oncol Biol Phys. 2012 Nov 15;84(4):943-8. doi: 10.1016/j.ijrobp.2012.01.067. Epub 2012 Apr 9. PMID 22494581
- [Background] Bentzen SM, Constine LS, Deasy JO, Eisbruch A, Jackson A, Marks LB, Ten Haken RK, Yorke ED. Quantitative Analyses of Normal Tissue Effects in the Clinic (QUANTEC): an introduction to the scientific issues. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3 Suppl):S3-9. doi: 10.1016/j.ijrobp.2009.09.040. PMID 20171515
- [Background] Lin NU, Lee EQ, Aoyama H, Barani IJ, Barboriak DP, Baumert BG, Bendszus M, Brown PD, Camidge DR, Chang SM, Dancey J, de Vries EG, Gaspar LE, Harris GJ, Hodi FS, Kalkanis SN, Linskey ME, Macdonald DR, Margolin K, Mehta MP, Schiff D, Soffietti R, Suh JH, van den Bent MJ, Vogelbaum MA, Wen PY; Response Assessment in Neuro-Oncology (RANO) group. Response assessment criteria for brain metastases: proposal from the RANO group. Lancet Oncol. 2015 Jun;16(6):e270-8. doi: 10.1016/S1470-2045(15)70057-4. Epub 2015 May 27. PMID 26065612
- [Background] Kocher M, Soffietti R, Abacioglu U, Villa S, Fauchon F, Baumert BG, Fariselli L, Tzuk-Shina T, Kortmann RD, Carrie C, Ben Hassel M, Kouri M, Valeinis E, van den Berge D, Collette S, Collette L, Mueller RP. Adjuvant whole-brain radiotherapy versus observation after radiosurgery or surgical resection of one to three cerebral metastases: results of the EORTC 22952-26001 study. J Clin Oncol. 2011 Jan 10;29(2):134-41. doi: 10.1200/JCO.2010.30.1655. Epub 2010 Nov 1. PMID 21041710
- [Derived] El Shafie RA, Paul A, Bernhardt D, Hauswald H, Welzel T, Sprave T, Hommertgen A, Krisam J, Schmitt D, Kluter S, Schubert K, Klose C, Kieser M, Debus J, Rieken S. Evaluation of Stereotactic Radiotherapy of the Resection Cavity After Surgery of Brain Metastases Compared to Postoperative Whole-Brain Radiotherapy (ESTRON)-A Single-Center Prospective Randomized Trial. Neurosurgery. 2018 Sep 1;83(3):566-573. doi: 10.1093/neuros/nyy021. PMID 29528419